CLINICAL TRIAL: NCT06444802
Title: Model-informed Precision Dosing for Linezolid: a Pilot Randomized Clinical Trial
Brief Title: Model-informed Precision Dosing for Linezolid
Acronym: LINEMAP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Flaminia Olearo, Principal Investigator, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTU 08.922
Record Dates: First submitted 2024-05-24; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: Linezolid; PK-PD Model; TDM
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linezolid Dosing based on TDMx (Experimental): Linezolid dosing based on a model-informed precision dosing (TDMx)
  Interventions: Drug: Linezolid
- Standard Linezolid dosing (Active Comparator): Patient will receive Linezolid at standard dose
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — Linezolid dosing will be adapted according to a model informed precision dosing (TDMx)

SUMMARY:
Study Rationale: Previous in vitro and retrospective in vivo studies suggest that optimal linezolid concentrations (between 2 and 7 mg/L) achieve clinical efficacy and microbiological eradication while minimizing side effects like thrombocytopenia and the emergence of resistance. No prospective or randomized clinical trial has confirmed these findings, and there is no consensus on how to adjust linezolid dosing to achieve optimal drug concentrations.

Objectives: The primary objective is to determine if model-informed precision dosing optimizes linezolid dosing to achieve therapeutic trough concentrations compared to a standard dose. Secondary objectives include assessing the PK/PD profile, investigating the prevalence of linezolid resistance among gram-positive bacteria, assessing microbiological resolution of infection, and evaluating the safety and tolerability of linezolid.

Methodology: This study is an open, monocentric pilot randomized controlled trial with two arms: standard dose therapy versus dose adjustment based on model-informed precision dosing using therapeutic drug monitoring and PK/PD targets developed in TMDx software.

Sample Size: 28 patients, 14 in each group. Assumptions are based on only 25% of patients in intensive care achieving the optimal therapeutic range with standard dosing, compared to an expected 80% achieving this with model-informed precision dosing.

Selection Criteria: Adult patients (18+ years) already starting linezolid treatment for gram-positive infections, expected to require treatment beyond the next calendar day. Exclusions include imminent death, expected or confirmed pregnancy, expected linezolid treatment of less than 4 days or more than 4 weeks.

Outcomes: The primary endpoint is defined as the difference in the proportion of patients in the intervention and in the control groups who maintained a trough linezolid concentration of 2 to 7 mg/L on Day 7 and Day 13.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Linezolid treatment is indicated or has been started due to pneumonia, skin or soft tissue infection; the patient has received no more than 2 infusions of 600 mg linezolid each
3. with written informed consent of the patient or
4. with written informed consent of his/her legal representative or
5. after using the option of inclusion via spouse according to § 1358 BGB or
6. after application of the independent consultant procedure
7. Patients of childbearing age: negative pregnancy test

Exclusion Criteria:

1. Patients receiving antibiotics active against Gram-positive bacteria at the same time of linezolid
2. Infection other than pneumonia, skin or soft tissue infection, especially tuberculosis, endocarditis and osteomyelitis
3. Death is deemed imminent and inevitable
4. Pregnancy
5. Lactation/breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Through concentration in the target | Day 7 of linezolid treatment
  The primary endpoint is defined as the likehood in achieving a trough linezolid concentration of 2 to 8 mg/L on Day 7

SECONDARY OUTCOMES:
Pharmacokinetic: | Day 7 and day 13 of linezolid treatment
  Percentage of the dosing interval while drug concentration remains above the MIC (f%T > MIC)
Thrombocytopenia | From the start of linezolid treatment and up to 14 days
  Median variation of platelets count after the start up to end of linezolid treatment
lactic acidosis and peripheral neuropathy | From the start of linezolid treatment and up to 14 days
  Frequency of lactic acidosis and peripheral neuropathy
Microbiology | From the start of linezolid treatment and up to 14 days
  Time to microbiologic eradication is calculated as the interval between the first isolation of a Gram-positive pathogen causing the infection and the first negative culture from the same type of biological material
Microbiology | From the start of linezolid treatment and up to 14 days
  Time to development of resistance to linezolid in Gram-positive bacteria is calculated as the interval in days between the first isolation of a specific bacteria species sensitive to linezolid and the first isolation of the same species showing resistance, in any type of biological material.
Microbiology | At the end of treatment up to the end of 30 day follow-up
  Rate of Relapse of gram-positive infection (growth of the same gram-positive organism in the blood culture or in another primarily site infected up to EOF).

IPD SHARING:
Plan to Share IPD: No